CLINICAL TRIAL: NCT02151422
Title: Breathing Exercises for Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Alan Baptist, MD, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00081294.
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Asthma
Keywords: Adults; age 18-65; physician-diagnosed; persistent asthma
MeSH Terms: conditions — Asthma | interventions — Breathing Exercises; Methods

ARMS (1):
- Breathing exercises (Experimental): Patients will be thought 3 different exercises included yoga pranayama, diaphragmatic breathing and pursed lip breathing. Patients will be asked to repeat these exercises at least twice daily for a one month period. Also patients will be thought 4 different exercises which they could use in the event of an asthma exacerbation. Teaching will be supplemented by a breathing exercise brochure and patients will be asked to demonstrate proper technique at initial visit and at the return visit.
  Interventions: Behavioral: Breathing exercise

INTERVENTIONS:
Behavioral: Breathing exercise — Patients will be thought 3 different exercises included yoga pranayama, diaphragmatic breathing and pursed lip breathing. Patients will be asked to repeat these exercises at least twice daily for a one month period. Also patients will be thought 4 different exercises which they could use in the event of an asthma exacerbation. Teaching will be supplemented by a breathing exercise brochure and patients will be asked to demonstrate proper technique at initial visit and at the return visit.
  Other Names: Intervention

SUMMARY:
Despite the advances in pharmacological therapy for asthma, there has been an increasing worldwide interest in alternative therapies for asthma. Treatments and therapies such as yoga, acupuncture, homeopathy, hypnosis and Buteyko and other breathing techniques have been used as complementary therapies however little evidence exists behind such practices.

Data from systemic reviews and randomized control trials provide evidence of benefit although additional confirmation is still needed. Among the most common techniques are the Buteyko breathing exercises that aim to reduce minute ventilation by instruct asthmatics patients to breathe shallowly and slowly through the nose. The second common technique is the Pranayama, or yoga breathing exercises which emphasizes deep respirations and exhalation prolongation.

Our goal is to assess the effectiveness of breathing exercises as a complementary therapy for asthma.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18-65 of either sex, with a physician-diagnosed history of persistent asthma.
* Access to internet

Exclusion Criteria:

* Subjects with history of COPD or any other lung disease, pregnant or lactating women, no access to internet and patients who cannot communicate in English.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-11; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Improvement of quality of life of asthmatic patients | equal or greater than 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Alan Baptist, MD, Study Director — University of Michigan
Locations (1):
- Allergy and Immunology Clinic at University of Michigan, Ann Arbor, Michigan, United States